CLINICAL TRIAL: NCT01978275
Title: Are Stimulating Catheters More Efficacy for Lumbar Plexus Block Compared With Traditional Non-stimulating Ones? A Randomized, Prospective, Blinded, up and Down Study.
Brief Title: Stimulating Catheter for Lumbar Plexus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, Medical Doctor, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IOGPGC02-13
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-12

CONDITIONS: Knee Arthritis Disease
Keywords: total knee arthroplasty; lumbar plexus block; stimulating catheters; peripheral nerve blocks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stimulating catheters group (Experimental): Lumbar plexus block performed through stimulating catheter
  Interventions: Device: stimulong 100, pajunk, germany
- nonstimulating catheters (Active Comparator): lumbar plexus block through nonstimulating catheters
  Interventions: Device: plexolong 100, pajunk, germany

INTERVENTIONS:
Device: stimulong 100, pajunk, germany — simulating catheter
  Arms: stimulating catheters group
Device: plexolong 100, pajunk, germany — nonstimulating catheter
  Arms: nonstimulating catheters

SUMMARY:
Stimulating catheters have been introduced to reduce the incidence of secondary failure after continuous peripheral nerve blocks, but they effectiveness over traditional nonstimulating catheters is still controversial. Furthermore no volume-response study has compared the success rates of the two techniques for continuous lumbar plexus block. The aim of this prospective, randomized, blinded study is to detect if stimulating catheters decrease the minimal effective volume (MEAV) of 1.5% mepivacaine required for successful lumbar plexus block (LPB) in 50% of patients compared with conventional non-stimulating catheters.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee arthroplasty

Exclusion Criteria:

* diabetes
* coagulation disorders
* allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
minimum effective anesthetic volume in 50% of patients | thirty minutes after local anesthetic injection

SECONDARY OUTCOMES:
morphine requirement | intraoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico G. Pini, Milan, Milano, Italy